CLINICAL TRIAL: NCT00107276
Title: Phase II Trial of Simple Oral Therapy (Continuous Oral Cyclophosphamide and Capecitabine) in Patients With Metastatic Breast Cancer
Brief Title: S0430 Cyclophosphamide and Capecitabine in Treating Women With Stage IV Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000423180; S0430 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2005-04-05; First posted 2005-04-06 (Estimated); Results first posted 2013-06-27 (Estimated); Last update posted 2013-07-18 (Estimated); Status verified 2013-07

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- cyclophosphamide and capecitabine (Experimental): cyclophosphamide orally days 1-14 and capecitabine orally days 15-21 for 8 cycles of 21 days each
  Interventions: Drug: capecitabine; Drug: cyclophosphamide

INTERVENTIONS:
Drug: capecitabine
Drug: cyclophosphamide
  Other Names: cytoxan

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as cyclophosphamide and capecitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one chemotherapy drug may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving cyclophosphamide together with capecitabine works in treating women with stage IV breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate (complete and partial, confirmed and unconfirmed) in women with stage IV breast cancer treated with oral cyclophosphamide and oral capecitabine.
* Determine the progression-free survival and overall survival of patients treated with this regimen.
* Determine the toxicity of this regimen in these patients.
* Determine the quality of life of patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive oral cyclophosphamide once daily on days 1-14 and oral capecitabine twice daily on days 8-21. Treatment repeats every 21 days for up to 8 courses in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline and then at weeks 7, 13, 19, and 25.

After completion of study treatment, patients are followed every 3 months for up to 2 years.

PROJECTED ACCRUAL: A total of 96 patients will be accrued for this study within 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed stage IV breast cancer

  * Metastatic disease (M1) OR multiple sites of new disease that is clinically obvious metastatic disease (i.e., multiple sites of new osseous disease)
* Meets 1 of the following criteria:

  * Measurable disease
  * Non-measurable disease

    * MUC-1 antigen level > 2 times upper limit of normal AND level has increased by 1.5 times
* Must have documented MUC-1 antigen level

  * Either cancer antigen (CA) 15-3 or CA 27-29 allowed
* Must have received at least 1 prior hormonal therapy for metastatic disease (estogen receptor-positive patients only)
* No symptomatic brain or CNS metastases

  * Previously treated brain or CNS metastasis allowed provided radiotherapy was completed ≥ 8 weeks before study entry
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Female

Menopausal status

* Not specified

Performance status

* Zubrod 0-2

Life expectancy

* Not specified

Hematopoietic

* No known existing uncontrolled coagulopathy

Hepatic

* Not specified

Renal

* Creatinine clearance > 40 mL/min

Cardiovascular

* No congestive heart failure
* No symptomatic coronary artery disease
* No cardiac arrhythmia not well controlled with medication
* No myocardial infarction within the past 12 months
* No other clinically significant cardiac disease

Gastrointestinal

* Able to take oral medication
* No uncontrolled nausea, vomiting, or diarrhea
* No lack of physical integrity of the upper gastrointestinal tract
* No malabsorption syndrome

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No active infection requiring systemic therapy
* No prior severe reaction to fluoropyrimidines
* No known sensitivity to fluorouracil
* No known dihydropyrimidine dehydrogenase deficiency
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent immunotherapy or biologic therapy for breast cancer
* No concurrent gene therapy for breast cancer
* No concurrent filgrastim (G-CSF)

Chemotherapy

* At least 14 days since prior chemotherapy and recovered
* No more than 2 prior chemotherapy regimens for metastatic disease
* No prior capecitabine for metastatic disease
* No prior oral cyclophosphamide for metastatic disease

  * Prior IV cyclophosphamide allowed
* No other concurrent chemotherapy for breast cancer

Endocrine therapy

* See Disease Characteristics
* No concurrent hormonal therapy for breast cancer

Radiotherapy

* See Disease Characteristics
* At least 14 days since prior radiotherapy to non-CNS disease sites and recovered
* No concurrent radiotherapy for breast cancer

Surgery

* Not specified

Other

* Concurrent bisphosphonates allowed
* No concurrent full-dose warfarin

  * Concurrent prophylactic warfarin (≤ 1 mg/day) to maintain port patency allowed
* No other concurrent antineoplastic therapy for breast cancer

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2005-08; Primary Completion 2008-03 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne F. Schott, MD, Study Chair — University of Michigan Rogel Cancer Center; Kathy S. Albain, MD, Study Chair — Loyola University
Locations (145):
- United States (145):
  - Alaska Regional Hospital Cancer Center, Anchorage, Alaska
  - Providence Cancer Center, Anchorage, Alaska
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Eden Medical Center, Castro Valley, California
  - Kaiser Permanente - Fremont, Fremont, California
  - Kaiser Permanente Medical Center - Hayward, Hayward, California
  - Saint Rose Hospital, Hayward, California
  - Highland General Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Kaiser Permanente Medical Center - Oakland, Oakland, California
  - Valley Care Medical Center, Pleasanton, California
  - Kaiser Permanente Medical Center - Redwood City, Redwood City, California
  - Kaiser Permanente Medical Center - Richmond, Richmond, California
  - Kaiser Permanente Medical Center - Roseville, Roseville, California
  - University of California Davis Cancer Center, Sacramento, California
  - South Sacramento Kaiser-Permanente Medical Center, Sacramento, California
  - Kaiser Permanente Medical Center - Sacramento, Sacramento, California
  - Kaiser Permanente Medical Center - San Francisco Geary Campus, San Francisco, California
  - Kaiser Permanente Medical Center - Santa Teresa, San Jose, California
  - Doctors Medical Center - San Pablo Campus, San Pablo, California
  - Kaiser Foundation Hospital - San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara Kiely Campus, Santa Clara, California
  - Kaiser Permanente Medical Center - Santa Rosa, Santa Rosa, California
  - Kaiser Permanente Medical Center - South San Francisco, South San Francisco, California
  - Kaiser Permanente Medical Facility - Stockton, Stockton, California
  - Kaiser Permanente Medical Center - Vallejo, Vallejo, California
  - Kaiser Permanente Medical Center - Walnut Creek, Walnut Creek, California
  - University of Colorado Cancer Center at UC Health Sciences Center, Aurora, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - Shaw Cancer Center at Vail Valley Medical Center, Edwards, Colorado
  - Curtis & Elizabeth Anderson Cancer Institute at Memorial Health University Medical Center, Savannah, Georgia
  - Pearlman Comprehensive Cancer Center at South Georgia Medical Center, Valdosta, Georgia
  - Saint Anthony's Hospital at Saint Anthony's Health Center, Alton, Illinois
  - Decatur Memorial Hospital Cancer Care Institute, Decatur, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Edward Hospital Cancer Center, Naperville, Illinois
  - Regional Cancer Center at Memorial Medical Center, Springfield, Illinois
  - Cancer Center of Kansas, PA - Chanute, Chanute, Kansas
  - Cancer Center of Kansas, PA - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas, PA - El Dorado, El Dorado, Kansas
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Cancer Center of Kansas, PA - Kingman, Kingman, Kansas
  - Southwest Medical Center, Liberal, Kansas
  - Cancer Center of Kansas, PA - Newton, Newton, Kansas
  - Cancer Center of Kansas, PA - Parsons, Parsons, Kansas
  - Cancer Center of Kansas, PA - Pratt, Pratt, Kansas
  - Cancer Center of Kansas, PA - Salina, Salina, Kansas
  - Tammy Walker Cancer Center at Salina Regional Health Center, Salina, Kansas
  - Cotton-O'Neil Cancer Center, Topeka, Kansas
  - St. Francis Comprehensive Cancer Center, Topeka, Kansas
  - Cancer Center of Kansas, PA - Wellington, Wellington, Kansas
  - Associates in Womens Health, PA - North Review, Wichita, Kansas
  - Cancer Center of Kansas, PA - Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas, PA - Wichita, Wichita, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Via Christi Cancer Center at Via Christi Regional Medical Center, Wichita, Kansas
  - Cancer Center of Kansas, PA - Winfield, Winfield, Kansas
  - Caritas Holy Family Hospital, Methuen, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Breslin Cancer Center at Ingham Regional Medical Center, Lansing, Michigan
  - Ted B. Wahby Cancer Center at Mount Clemens General Hospital, Mount Clemens, Michigan
  - William Beaumont Hospital - Royal Oak Campus, Royal Oak, Michigan
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Southeast Missouri Regional Cancer Center at Southeast Missouri Hospital, Gape Girardeau, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - Saint Louis University Cancer Center, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - David C. Pratt Cancer Center at St. John's Mercy, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare Cancer Care Services, Billings, Montana
  - Billings Clinic - Downtown, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - St. James Healthcare Cancer Care, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic - Main Facility, Great Falls, Montana
  - Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology at KRMC, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Center, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Adirondack Cancer Care - Glens Falls, Glens Falls, New York
  - Wayne Memorial Hospital, Incorporated, Goldsboro, North Carolina
  - Iredell Memorial Hospital, Statesville, North Carolina
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Community Oncology Group at Cleveland Clinic Cancer Center, Independence, Ohio
  - MedCentral - Mansfield Hospital, Mansfield, Ohio
  - Cleveland Clinic - Wooster, Wooster, Ohio
  - Legacy Mount Hood Medical Center, Gresham, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Legacy Good Samaritan Hospital & Medical Center Comprehensive Cancer Center, Portland, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Legacy Emanuel Hospital and Health Center & Children's Hospital, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Roper St. Francis Cancer Center at Roper Hospital, Charleston, South Carolina
  - Center for Cancer Medicine and Blood Disorders, PA, El Paso, Texas
  - American Fork Hospital, American Fork, Utah
  - Sandra L. Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Cottonwood Hospital Medical Center, Murray, Utah
  - Jon and Karen Huntsman Cancer Center at Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center - Provo, Provo, Utah
  - Latter Day Saints Hospital, Salt Lake City, Utah
  - Utah Cancer Specialists at UCS Cancer Center, Salt Lake City, Utah
  - Dixie Regional Medical Center - East Campus, St. George, Utah
  - Auburn Regional Center for Cancer Care, Auburn, Washington
  - St. Joseph Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Providence Centralia Hospital, Centralia, Washington
  - St. Francis Hospital, Federal Way, Washington
  - Skagit Valley Hospital Cancer Care Center, Mount Vernon, Washington
  - Providence St. Peter Hospital Regional Cancer Center, Olympia, Washington
  - Good Samaritan Cancer Center, Puyallup, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Minor and James Medical, PLLC, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - Polyclinic First Hill, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - St. Joseph Medical Center at Franciscan Health System, Tacoma, Washington
  - Allenmore Hospital, Tacoma, Washington
  - CCOP - Northwest, Tacoma, Washington
  - MultiCare Regional Cancer Center at Tacoma General Hospital, Tacoma, Washington
  - St. Clare Hospital, Tacoma, Washington
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington
  - United Hospital Center, Clarksburg, West Virginia
  - Community Comprehensive Cancer Center at Camden-Clark Memorial Hospital, Parkersburg, West Virginia
  - Welch Cancer Center at Sheridan Memorial Hospital, Sheridan, Wyoming

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between 8/15/2005 and 9/1/2007, 112 patients were registered from 26 SWOG institutions who obtained Institutional Review Board (IRB) approval for the study.
Period: Overall Study
Arm/Group | Cyclophosphamide and Capecitabine
Started | 112
Eligible | 96
Completed | 40
Not Completed | 72
Not completed — Progression | 46
Not completed — Adverse Event | 6
Not completed — M.D. decision | 2
Not completed — Patient refusal | 1
Not completed — Death | 1
Not completed — Ineligible | 16

BASELINE CHARACTERISTICS:
Arm/Group | Cyclophosphamide and Capecitabine
Number analyzed (Participants) | 96
Age Continuous [Median (Full Range); unit: years] | 59.7 [34.3 to 88.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Response Rate (Complete and Partial, Confirmed and Unconfirmed)
Description: Complete Response (CR) is complete disappearance of all measurable and non-measurable disease. No new lesions, no disease related symptoms. Normalization of markers and other abnormal lab values. Partial Response (PR) is greater than or equal to 30% decrease under baseline of the sum of longest diameters of all target measurable lesions. No unequivocal progression of non-measurable disease. No new lesions. Confirmation of CR or PR means a repeat scan at least 4 weeks apart documented before progression or symptomatic deterioration. Progression is 20% increase in sum of longest diameters of target measurable lesions over smallest sum observed and/or unequivocal progression of non-measurable disease and/or appearance of new lesion/site or death due to disease without prior documentation of progression and without symptomatic deterioration. Symptomatic deterioration is global deterioration of health status requiring discontinuation of treatment without objective evidence of progression.
Time Frame: Patients assessed at least every six weeks while on protocol treatment
Population: Eligible patients with RECIST measurable disease
Measure: Number; unit: participants
Arm/Group | Cyclophosphamide and Capecitabine
Number analyzed (Participants) | 80
participants | 29 [26% to 48%]

2. Secondary Outcome: Progression-free Survival and Overall Survival
Description: Progression-Free Survival: From date of registration to time of first documentation of progression or symptomatic deterioration, or death due to any cause. Patients last known to be alive and progression-free are censored at last date of contact.
  Overall Survival: From date of registration to date of death due to any cause. Patients last known to be alive are censored at last date of contact.
  Progression is 20% increase in sum of longest diameters of target measurable lesions over smallest sum observed and/or unequivocal progression of non-measurable disease and/or appearance of new lesion/site or death due to disease without prior documentation of progression and without symptomatic deterioration. Symptomatic deterioration is global deterioration of health status requiring discontinuation of treatment without objective evidence of progression.
Time Frame: two years
Population: All eligible patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cyclophosphamide and Capecitabine
Number analyzed (Participants) | 96
months
  PFS | 5.9 [3.7 to 8.0]
  OS | 18.8 [13.1 to 22.0]

3. Secondary Outcome: Toxicity
Description: Number of patients for whom Grade 3 or higher toxicity observed during treatment. Only adverse events that are possibly, probably or definitely related to study drug are reported.
Time Frame: Patients assessed after each 21-day cycle for 8 cycles (24 weeks of treatment)
Population: Eligible patients evaluable for toxicity assessment (one eligible patient who was removed from treatment due to disease progression less than 3 weeks after registration is not evaluable for toxicity assessment)
Measure: Number; unit: Participants
Arm/Group | Cyclophosphamide and Capecitabine
Number analyzed (Participants) | 95
Participants
  ALT, SGPT (serum glutamic pyruvic transaminase) | 1
  Alkaline phosphatase | 1
  Dehydration | 2
  Diarrhea | 2
  Dyspnea (shortness of breath) | 1
  Fatigue (asthenia, lethargy, malaise) | 2
  Febrile neutropenia | 1
  Hemoglobin | 1
  Leukocytes (total WBC) | 15
  Lymphopenia | 13
  Mood alteration - depression | 1
  Nausea | 1
  Neuroendocrine: ADH secretion abnormality | 1
  Neutrophils/granulocytes (ANC/AGC) | 7
  Platelets | 1
  Potassium, serum-low (hypokalemia) | 1
  Pruritus/itching | 1
  Rash/desquamation | 1
  Rash: hand-foot skin reaction | 7
  Sodium, serum-low (hyponatremia) | 1
  Thrombosis/thrombus/embolism | 2
  Weight loss | 1

ADVERSE EVENTS:
Time Frame: Every 3 weeks for up to 2 years.
Description: Number "At Risk" includes all eligible patients evaluable for toxicity assessment (one eligible patient who was removed from treatment due to disease progression less than 3 weeks after registration is not evaluable for toxicity assessment)
Arm/Group | Cyclophosphamide and Capecitabine
Serious Adverse Events (participants affected / at risk) | 4/95
Other Adverse Events (participants affected / at risk) | 92/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cyclophosphamide and Capecitabine (N=95)
Death not associated with CTCAE term - Death NOS (General disorders) | 1
Death - Disease progression NOS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
CNS cerebrovascular ischemia (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cyclophosphamide and Capecitabine (N=95)
Hemoglobin (Blood and lymphatic system disorders) | 40
Constipation (Gastrointestinal disorders) | 16
Diarrhea (Gastrointestinal disorders) | 32
Heartburn/dyspepsia (Gastrointestinal disorders) | 10
Mucositis/stomatitis (clinical exam) - Oral cavity (Gastrointestinal disorders) | 8
Mucositis/stomatitis (functional/symp) - Oral cav (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 53
Pain - Abdomen NOS (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 28
Edema: limb (General disorders) | 11
Fatigue (asthenia, lethargy, malaise) (General disorders) | 61
Pain-Other (Specify) (General disorders) | 10
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 12
AST, SGOT (Investigations) | 18
Alkaline phosphatase (Investigations) | 19
Bilirubin (hyperbilirubinemia) (Investigations) | 11
Leukocytes (total WBC) (Investigations) | 43
Lymphopenia (Investigations) | 21
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 29
Platelets (Investigations) | 13
Weight loss (Investigations) | 8
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 5
Anorexia (Metabolism and nutrition disorders) | 23
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 7
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 29
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 8
Sodium, serum-low (hyponatremia) (Metabolism and nutrition disorders) | 12
Muscle weakness, not d/t neuropathy - body/general (Musculoskeletal and connective tissue disorders) | 5
Pain - Back (Musculoskeletal and connective tissue disorders) | 10
Pain - Bone (Musculoskeletal and connective tissue disorders) | 13
Pain - Extremity-limb (Musculoskeletal and connective tissue disorders) | 8
Pain - Joint (Musculoskeletal and connective tissue disorders) | 7
Dizziness (Nervous system disorders) | 12
Neuropathy: sensory (Nervous system disorders) | 14
Pain - Head/headache (Nervous system disorders) | 8
Taste alteration (dysgeusia) (Nervous system disorders) | 9
Insomnia (Psychiatric disorders) | 6
Mood alteration - anxiety (Psychiatric disorders) | 11
Mood alteration - depression (Psychiatric disorders) | 15
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 10
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 20
Dry skin (Skin and subcutaneous tissue disorders) | 7
Hair loss/Alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 5
Nail changes (Skin and subcutaneous tissue disorders) | 7
Rash/desquamation (Skin and subcutaneous tissue disorders) | 5
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 37
Hot flashes/flushes (Vascular disorders) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No